CLINICAL TRIAL: NCT00168831
Title: A Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Efficacy and Safety Comparison of One-Year Treatment of Two Doses (5mg and 10mg) of Tiotropium Inhalation Solution Delivered by the Respimat Device in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Tiotropium / Respimat One-Year Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.255
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2009-10-07 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2013-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (3):
- Tiotropium Respimat 5mcg (Tio R5) (Other)
  Interventions: Drug: Tiotropium Inhalation Solution
- Tiotropium Respimat 10mcg (Tio R10) (Other)
  Interventions: Drug: Tiotropium Inhalation Solution
- Placebo (Other)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tiotropium Inhalation Solution
  Arms: Tiotropium Respimat 10mcg (Tio R10); Tiotropium Respimat 5mcg (Tio R5)
Other: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the long term effects of treatment with two doses of Tiotropium delivered by the Respimat inhaler in patients with COPD.

ELIGIBILITY:
Criteria

* Patients with stable moderate to severe COPD and a smoking history of at least 10 pack years were eligible for inclusion in the study. Patients with significant diseases other than COPD were excluded as were patients with a recent history of myocardial infarction, history of malignancy, unstable or life-threatening cardiac arrhythmia, narrow-angle glaucoma, asthma or other allergic conditions. Patients treated with cromolyn, nedocromil, oral beta-adrenergics or unstable doses of oral corticosteroids were ineligible for inclusion in the study as were patients who had received previous treatment with tiotropium.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1007 (Actual)
Dates: Start 2003-02; Primary Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (76):
- United States (12):
  - Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - Boehringer Ingelheim Investigational Site, La Jolla, California
  - Boehringer Ingelheim Investigational Site, Long Beach, California
  - Boehringer Ingelheim Investigational Site, San Luis Obispo, California
  - Boehringer Ingelheim Investigational Site, Gainesville, Florida
  - Boehringer Ingelheim Investigational Site, Hallandale, Florida
  - Boehringer Ingelheim Investigational Site, Hines, Illinois
  - Boehringer Ingelheim Investigational Site, Chesterfield, Missouri
  - Boehringer Ingelheim Investigational Site, Bay Shore, New York
  - Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - Boehringer Ingelheim Investigational Site, Houston, Texas
  - Boehringer Ingelheim Investigational Site, Richmond, Virginia
- Australia (3):
  - Boehringer Ingelheim Investigational Site, Garran, Australian Capital Territory
  - Boehringer Ingelheim Investigational Site, Adelaide, South Australia
  - Boehringer Ingelheim Investigational Site, Nedlands, Western Australia
- Austria (6):
  - Boehringer Ingelheim Investigational Site, Innsbruck
  - Boehringer Ingelheim Investigational Site, Mittersill
  - Boehringer Ingelheim Investigational Site, Schwechat
  - Baumgartner Hohe Otto Wagner Spital Wien, Vienna
  - Boehringer Ingelheim Investigational Site, Vienna
  - Boehringer Ingelheim Investigational Site, Wels
- Canada (5):
  - Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
- Finland (5):
  - Boehringer Ingelheim Investigational Site, Espoo
  - Boehringer Ingelheim Investigational Site, Helsinki
  - Boehringer Ingelheim Investigational Site, Lahti
  - Boehringer Ingelheim Investigational Site, Lappeenranta
  - Boehringer Ingelheim Investigational Site, Lohja
- France (6):
  - Boehringer Ingelheim Investigational Site, Amboise
  - Boehringer Ingelheim Investigational Site, Chauny
  - Boehringer Ingelheim Investigational Site, Marseille
  - Boehringer Ingelheim Investigational Site, Metz
  - Boehringer Ingelheim Investigational Site, Montpellier
  - Boehringer Ingelheim Investigational Site, Nantes
- Greece (4):
  - Boehringer Ingelheim Investigational Site, Alexandroupoli
  - Boehringer Ingelheim Investigational Site, Athens
  - Boehringer Ingelheim Investigational Site, Mournies-Chania
  - Boehringer Ingelheim Investigational Site, Trikala
- Boehringer Ingelheim Investigational Site, Dublin, Ireland
- Italy (10):
  - Boehringer Ingelheim Investigational Site, Bologna
  - Boehringer Ingelheim Investigational Site, Bussolengo (vr)
  - Boehringer Ingelheim Investigational Site, Cava Dei Tirreni (SA)
  - Boehringer Ingelheim Investigational Site, Crema (CR)
  - Boehringer Ingelheim Investigational Site, Genova
  - Boehringer Ingelheim Investigational Site, Milan
  - Boehringer Ingelheim Investigational Site, Pistoia
  - Boehringer Ingelheim Investigational Site, Roma
  - Boehringer Ingelheim Investigational Site, Salerno
  - Boehringer Ingelheim Investigational Site, Sesto San Giovanni (Milano)
- Netherlands (6):
  - Boehringer Ingelheim Investigational Site, Arnhem
  - Boehringer Ingelheim Investigational Site, Eindhoven
  - Boehringer Ingelheim Investigational Site, Heerenveen
  - Boehringer Ingelheim Investigational Site, Hoorn
  - Boehringer Ingelheim Investigational Site, Leeuwarden
  - Boehringer Ingelheim Investigational Site, Rotterdam
- New Zealand (2):
  - Boehringer Ingelheim Investigational Site, Auckland
  - Boehringer Ingelheim Investigational Site, Hamilton
- Boehringer Ingelheim Investigational Site, Saint Petersburg, Russia
- South Africa (5):
  - Boehringer Ingelheim Investigational Site, Bellville
  - Boehringer Ingelheim Investigational Site, Cape Town
  - Boehringer Ingelheim Investigational Site, George
  - Boehringer Ingelheim Investigational Site, Johannesburg
  - Boehringer Ingelheim Investigational Site, Vanderbijlpark
- Spain (4):
  - Boehringer Ingelheim Investigational Site, Barcelona
  - Boehringer Ingelheim Investigational Site, Centelles
  - Boehringer Ingelheim Investigational Site, Murcia
  - Boehringer Ingelheim Investigational Site, Sant Boi de Llobregat (Barcelona)
- United Kingdom (6):
  - Boehringer Ingelheim Investigational Site, Babbacombe
  - Boehringer Ingelheim Investigational Site, Cottingham
  - Boehringer Ingelheim Investigational Site, Isleworth
  - Boehringer Ingelheim Investigational Site, Manchester
  - Boehringer Ingelheim Investigational Site, Plymouth
  - Boehringer Ingelheim Investigational Site, Sunderland

REFERENCES:
- [Derived] Singh D, Wedzicha JA, Siddiqui S, de la Hoz A, Xue W, Magnussen H, Miravitlles M, Chalmers JD, Calverley PMA. Blood eosinophils as a biomarker of future COPD exacerbation risk: pooled data from 11 clinical trials. Respir Res. 2020 Sep 17;21(1):240. doi: 10.1186/s12931-020-01482-1. PMID 32943047
- [Derived] Hohlfeld JM, Furtwaengler A, Konen-Bergmann M, Wallenstein G, Walter B, Bateman ED. Cardiac safety of tiotropium in patients with COPD: a combined analysis of Holter-ECG data from four randomised clinical trials. Int J Clin Pract. 2015 Jan;69(1):72-80. doi: 10.1111/ijcp.12596. Epub 2014 Dec 11. PMID 25496316
- [Derived] Hodder R, Pavia D, Lee A, Bateman E. Lack of paradoxical bronchoconstriction after administration of tiotropium via Respimat(R) Soft Mist Inhaler in COPD. Int J Chron Obstruct Pulmon Dis. 2011;6:245-51. doi: 10.2147/COPD.S16094. Epub 2011 Apr 26. PMID 21814460

RESULTS

PARTICIPANT FLOW:
Groups:
- Tiotropium Respimat 5mcg (Tio R5): Tiotropium Bromide inhalation solution delivered from Respimat Inhaler (5 mcg)
- Tiotropium Respimat 10mcg (Tio R10): Tiotropium Bromide inhalation solution delivered from Respimat Inhaler (10 mcg)
- Placebo: Placebo inhalation solution delivered from Respimat Inhaler (matching placebo)
Period: Overall Study
Arm/Group | Tiotropium Respimat 5mcg (Tio R5) | Tiotropium Respimat 10mcg (Tio R10) | Placebo
Started | 338 | 335 | 334
Completed | 278 | 254 | 220
Not Completed | 60 | 81 | 114
Not completed — Adverse Event | 36 | 47 | 74
Not completed — Lost to Follow-up | 5 | 6 | 4
Not completed — Withdrawal by Subject | 7 | 14 | 19
Not completed — Protocol Violation | 6 | 11 | 11
Not completed — Other | 6 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Tiotropium Respimat 5mcg: Tiotropium Bromide inhalation solution delivered from Respimat Inhaler (5 mcg)
- Tiotropium Respimat 10mcg: Tiotropium Bromide inhalation solution delivered from Respimat Inhaler (10 mcg)
- Total: Total of all reporting groups
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo | Total
Number analyzed (Participants) | 338 | 335 | 334 | 1007
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (8.9) | 65.6 (8.6) | 65.7 (8.4) | 65.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 89 | 99 | 278
  Male | 248 | 246 | 235 | 729

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough FEV1 After 48 Weeks
Description: Change From Baseline in Trough Forced Expiratory Volume in 1 second (FEV1) after 48 weeks
Time Frame: 10 minutes prior to test-drug inhalation and at 5, 30 and 60 minutes and 2 and 3 hours after inhalation of study medication
Population: Full Analysis Set - Clinic Spirometry (FAS-PFT)
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 324 | 324 | 307
Litres | 0.077 (0.012) | 0.105 (0.012) | -0.036 (0.012)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry, centre and baseline value; Mean Difference (Final Values) = 0.113, Standard Error of Mean 0.017 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry,centre and baseline value; Mean Difference (Final Values) = 0.140, Standard Error of Mean 0.017 — Tiotropium Respimat 10mcg - Placebo

2. Primary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score, Full Analysis Set - Saint George's Respiratory Questionnaire (FAS-QOL)
Description: Rating scale of 3 domains - symptoms, activities and impact (weighted). Worst score = 100, best score = 0
Time Frame: Week 48
Population: Full Analysis Set - Saint George's Respiratory Questionnaire (FAS-QOL)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 310 | 304 | 276
Points on a scale | 39.771 (0.718) | 40.038 (0.726) | 43.484 (0.763)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Test type: Superiority or Other; p = 0.0004, ANCOVA; The means are adjusted for centre, smoking status at entry and baseline value; Mean Difference (Final Values) = -3.713, Standard Error of Mean 1.052 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Test type: Superiority or Other; p = 0.0012, ANCOVA; The means are adjusted for centre, smoking status at entry and baseline value; Mean Difference (Final Values) = -3.445, Standard Error of Mean 1.059 — Tiotropium Respimat 10mcg - Placebo

3. Primary Outcome: TDI Focal Score, Full Analysis Set - Transitional Dyspnoea Index (FAS-TDI) (Combined Studies)
Description: Rating scale of 3 components - change in functional impairment, change in magnitude of tasks, change in magnitude of efforts. Worst score = -9, best score = +9
  For this endpoint data of twin studies NCT00168844 and NCT00168831 was combined.
Time Frame: Week 48
Population: Full Analysis Set - Transitional Dyspnoea Index (FAS-TDI)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 628 | 618 | 552
Points on a scale | 1.890 (0.112) | 1.913 (0.113) | 0.837 (0.120)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The means are adjusted for centre, smoking status at entry and baseline value; Mean Difference (Final Values) = 1.053, Standard Error of Mean 0.165 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The means are adjusted for centre, smoking status at entry and baseline value; Mean Difference (Final Values) = 1.075, Standard Error of Mean 0.166 — Tiotropium Respimat 10mcg - Placebo

4. Primary Outcome: COPD Exacerbation Rate, Safety Set (SS) (Combined Studies)
Description: Number of Chronic Obstructive Pulmonary Disease (COPD) exacerbations per patient year
  For this endpoint data of the twin studies NCT00168844 and NCT00168831 was combined.
Time Frame: 48 weeks
Population: Safety Set. Combined analysis of studies NCT00168844 and NCT00168831. 670 patients analysed in total comprises 338 patients from NCT00168831 and 332 patients from study NCT00168844, 667 patients - 335 and 332, 653 patients - 334 and 319 respectively.
Measure: Mean (Standard Deviation); unit: Number of exacerbations per patient year
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 670 | 667 | 653
Number of exacerbations per patient year | 0.93 (2.02) | 1.02 (3.05) | 1.91 (8.17)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Test type: Superiority or Other; p = 0.0002, Poisson regression; Odds Ratio (OR) = 0.782, 95% CI 2-sided [0.687 to 0.890] — Tiotropium Respimat 5mcg vs. Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Test type: Superiority or Other; p < 0.0001, Poisson regression; Odds Ratio (OR) = 0.725, 95% CI 2-sided [0.635 to 0.828] — Tiotropium Respimat 10mcg vs. Placebo

5. Secondary Outcome: Change From Baseline in Heart Rate
Description: Week 40 pre-dose - baseline
Time Frame: Baseline to Week 40 pre-dose
Population: Combined analysis of studies NCT00168844 and NCT00168831 in subset of patients who had additional 12-lead electrocardiogram (ECG) and 24-hour Holter monitoring performed (see protocol and clinical trial report)
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 155 | 135 | 109
beats per minute (bpm) | 2.1 (12.4) | 3.6 (10.5) | 1.8 (9.7)

6. Secondary Outcome: Change From Baseline in PR Interval
Time Frame: Baseline to Week 40 pre-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 150 | 131 | 105
milliseconds (msec) | -0.8 (20.2) | -2.5 (15.1) | -0.5 (15.3)

7. Secondary Outcome: Change From Baseline in QRS Interval
Description: Week 40 pre-dose - baseline
Time Frame: Baseline to Week 40 pre-dose
Population: Combined analysis of studies NCT00168844 and NCT00168831 in subset of patients who had additional 12-lead ECG and 24-hour Holter monitoring performed (see protocol and clinical trial report)
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 155 | 135 | 109
msec | 0.9 (9.4) | 1.7 (12.1) | -1.1 (10.3)

8. Secondary Outcome: Change From Baseline in QT Interval
Description: Week 40 pre-dose - baseline
Time Frame: Baseline to Week 40 pre-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 155 | 135 | 109
msec | -4.6 (26.5) | -3.5 (25.2) | -3.2 (22.3)

9. Secondary Outcome: Change From Baseline in QT Interval (Bazett)
Description: Week 40 pre-dose - baseline
Time Frame: Baseline to Week 40 pre-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 155 | 135 | 109
msec | -0.5 (29.9) | 5.4 (24.0) | 2.5 (23.4)

10. Secondary Outcome: Change From Baseline in QT Interval (Fridericia)
Description: Week 40 pre-dose - baseline
Time Frame: Baseline to Week 40 pre-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 155 | 135 | 109
msec | -2.0 (24.3) | 2.2 (21.3) | 0.5 (19.5)

11. Secondary Outcome: Change From Baseline in Heart Rate
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
bpm | 0.3 (5.4) | 1.2 (6.4) | 0.3 (6.6)

12. Secondary Outcome: Change From Baseline in Supraventricular Premature Beat (SVPB) Total
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: premature beats per 24 hours
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
premature beats per 24 hours | -3.4 (94.2) | 6.8 (87.4) | 20.9 (125.8)

13. Secondary Outcome: Change From Baseline in SVPB Run Events
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: events per 24 hours
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
events per 24 hours | 0.0 (0.6) | -0.1 (0.5) | -0.1 (1.6)

14. Secondary Outcome: Change From Baseline in SVPB Pairs
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pairs per 24 hours
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
pairs per 24 hours | -0.4 (4.0) | -0.2 (2.3) | 2.0 (16.4)

15. Secondary Outcome: Change From Baseline in Ventricular Premature Beat (VPB) Total
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: premature beats per 24 hours
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
premature beats per 24 hours | -14.3 (105.9) | 4.6 (68.8) | -24.1 (182.3)

16. Secondary Outcome: Change From Baseline in Ventricular Premature Beat (VPB) Run Events
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: events per 24 hours
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
events per 24 hours | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.0)

17. Secondary Outcome: Change From Baseline in VPB Pairs
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pairs per 24 hours
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
pairs per 24 hours | -0.2 (1.6) | -0.1 (3.8) | -0.9 (5.7)

18. Secondary Outcome: Change From Baseline in Haematocrit, Packed Cell Volume (PCV)
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: Percentage of erythrocytes
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 289 | 274 | 268
Percentage of erythrocytes | 0 (4) | 0 (4) | 0 (4)

19. Secondary Outcome: Change From Baseline in Haemoglobin
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: grams per litre (g/L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 299 | 280 | 276
grams per litre (g/L) | 0 (11) | -1 (10) | -1 (12)

20. Secondary Outcome: Change From Baseline in Red Blood Cell Count
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^12/Litre (L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 298 | 279 | 275
10^12/Litre (L) | 0.0 (0.3) | 0.0 (0.3) | 0.0 (0.3)

21. Secondary Outcome: Change From Baseline in White Blood Cell Count
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/Litre (L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 299 | 280 | 276
10^9/Litre (L) | 0.2 (1.7) | 0.3 (1.5) | 0.2 (1.5)

22. Secondary Outcome: Change From Baseline in Platelets
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 292 | 274 | 272
10^9/L | 5 (31) | 3 (29) | 0 (35)

23. Secondary Outcome: Change From Baseline in Neutrophils
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: percentage of white blood cell count
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 296 | 276 | 274
percentage of white blood cell count | 1 (8) | 1 (8) | 0 (8)

24. Secondary Outcome: Change From Baseline in Eosinophils
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: percentage of white blood cell count
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 296 | 276 | 274
percentage of white blood cell count | 0 (2) | 0 (2) | 0 (2)

25. Secondary Outcome: Change From Baseline in Basophils
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: percentage of white blood cell count
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 296 | 276 | 274
percentage of white blood cell count | 0 (0) | 0 (0) | 0 (0)

26. Secondary Outcome: Change From Baseline in Lymphocytes
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: percentage of white blood cell count
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 296 | 276 | 274
percentage of white blood cell count | -1 (4) | -1 (4) | 0 (4)

27. Secondary Outcome: Change From Baseline in Monocytes
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: percentage of white blood cell count
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 296 | 276 | 274
percentage of white blood cell count | 0 (4) | 0 (4) | 0 (4)

28. Secondary Outcome: Change From Baseline in Neutrophils (Absolute)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 296 | 276 | 274
10^9/L | 0.2 (1.9) | 0.3 (1.6) | 0.2 (1.6)

29. Secondary Outcome: Change From Baseline in Eosinophils (Absolute)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 296 | 276 | 274
10^9/L | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1)

30. Secondary Outcome: Change From Baseline in Basophils (Absolute)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 296 | 276 | 274
10^9/L | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1)

31. Secondary Outcome: Change From Baseline in Lymphocytes (Absolute)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 296 | 276 | 274
10^9/L | -0.1 (0.6) | 0.0 (0.7) | 0.0 (0.7)

32. Secondary Outcome: Change From Baseline in Monocytes (Absolute)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 296 | 276 | 274
10^9/L | 0.0 (0.3) | 0.0 (0.3) | 0.0 (0.3)

33. Secondary Outcome: Change From Baseline in Calcium
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: millimoles per litre (mmol/L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 304 | 284 | 277
millimoles per litre (mmol/L) | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.2)

34. Secondary Outcome: Change From Baseline in Phosphate
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 304 | 284 | 277
mmol/L | 0.01 (0.23) | 0.00 (0.24) | 0.02 (0.26)

35. Secondary Outcome: Change From Baseline in Aspartate Transaminase/Glutamic-oxaloacetic Transaminase (AST/GOT), Serum Glutamic-oxaloacetic Transaminase (SGOT)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: Units per litre (U/L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 304 | 284 | 277
Units per litre (U/L) | -1 (20) | -1 (25) | -2 (13)

36. Secondary Outcome: Change From Baseline in Alanine Transaminase/Glutamic Pyruvate Transaminase (ALT/GPT), Serum Glutamate Pyruvate Transaminase (SGPT)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 304 | 284 | 277
U/L | -1 (18) | -1 (18) | -1 (13)

37. Secondary Outcome: Change From Baseline in Alkaline Phosphatase
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 304 | 284 | 277
U/L | -4 (19) | -5 (23) | -3 (27)

38. Secondary Outcome: Change From Baseline in Lactic Dehyrogenase (LDH)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 302 | 282 | 276
U/L | 1 (40) | 3 (44) | 5 (42)

39. Secondary Outcome: Change From Baseline in Glucose
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 303 | 280 | 276
mmol/L | 0.02 (2.11) | 0.26 (2.17) | 0.10 (2.34)

40. Secondary Outcome: Change From Baseline in Urea
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 304 | 284 | 277
mmol/L | -0.2 (1.9) | 0.0 (2.1) | 0.1 (2.2)

41. Secondary Outcome: Change From Baseline in Blood Urea Nitrogen
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: milligrams per decilitre (mg/dL)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 304 | 284 | 277
milligrams per decilitre (mg/dL) | -0.3 (3.0) | 0.0 (3.3) | 0.2 (3.5)

42. Secondary Outcome: Change From Baseline in Creatinine
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: micromoles per litre (umol/L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 304 | 284 | 277
micromoles per litre (umol/L) | 2.2 (9.3) | 1.5 (12.2) | 2.1 (10.5)

43. Secondary Outcome: Change From Baseline in Bilirubin, Total
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 304 | 284 | 277
umol/L | -0.2 (5.2) | 0.4 (4.2) | -0.1 (4.6)

44. Secondary Outcome: Change From Baseline in Uric Acid
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 304 | 284 | 277
umol/L | 16.41 (80.08) | 9.39 (85.92) | 6.52 (76.49)

45. Secondary Outcome: Change From Baseline in Protein, Total
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: grams per litre (g/L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 304 | 284 | 277
grams per litre (g/L) | -1 (5) | -1 (5) | -1 (6)

46. Secondary Outcome: Change From Baseline in Albumin
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 304 | 284 | 277
g/L | 1 (4) | 1 (4) | 1 (4)

47. Secondary Outcome: Change From Baseline in Trough FEV1 After 2, 8, 16, 24, 32 and 40 Weeks
Description: Change From Baseline in Trough Forced Expiratory Volume in 1 second (FEV1) after 2, 8, 16, 24, 32 and 40 weeks. The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: as for outcome 1
Population: Full Analysis Set - Clinic Spirometry (FAS-PFT)
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 324 | 324 | 307
Litres
  Week 2 | 0.111 (0.010) | 0.114 (0.010) | -0.003 (0.011)
  Week 8 | 0.099 (0.011) | 0.133 (0.011) | -0.012 (0.011)
  Week 16 | 0.118 (0.012) | 0.132 (0.012) | -0.008 (0.012)
  Week 24 | 0.104 (0.012) | 0.132 (0.012) | -0.010 (0.012)
  Week 32 | 0.095 (0.012) | 0.145 (0.012) | -0.012 (0.013)
  Week 40 | 0.091 (0.012) | 0.106 (0.012) | -0.027 (0.012)

48. Secondary Outcome: Change From Baseline in Trough FVC After 2, 8, 16, 24, 32, 40 and 48 Weeks
Description: Change From Baseline in Trough Forced vital capacity (FVC) after 2, 8, 16, 24, 32, 40 and 48 weeks. The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: as for outcome 1
Population: Full Analysis Set - Clinic Spirometry (FAS-PFT)
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 324 | 324 | 307
Litres
  Week 2 | 0.257 (0.021) | 0.264 (0.022) | 0.009 (0.022)
  Week 8 | 0.207 (0.023) | 0.266 (0.023) | -0.007 (0.024)
  Week 16 | 0.259 (0.025) | 0.266 (0.025) | -0.002 (0.025)
  Week 24 | 0.236 (0.025) | 0.274 (0.025) | 0.008 (0.025)
  Week 32 | 0.203 (0.026) | 0.286 (0.026) | -0.008 (0.027)
  Week 40 | 0.211 (0.025) | 0.207 (0.025) | -0.028 (0.026)
  Week 48 | 0.197 (0.026) | 0.209 (0.026) | -0.043 (0.026)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry, centre and baseline value; Mean Difference (Final Values) = 0.240, Standard Error of Mean 0.037 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.252, Standard Error of Mean 0.037 — Tiotropium Respimat 10mcg - Placebo

49. Secondary Outcome: Change From Baseline in FEV1 AUC0-3 After 2, 8, 16, 24, 32, 40 and 48 Weeks
Description: FEV1 AUC0-3 represents the Area under Curve over the time interval from 0 to 3 hours after 2, 8, 16, 24, 32, 40 and 48 weeks. The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: as for outcome 1
Population: Full Analysis Set - Clinic Spirometry (FAS-PFT)
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 324 | 324 | 307
Litres
  Week 2 | 0.246 (0.011) | 0.257 (0.011) | 0.044 (0.012)
  Week 8 | 0.234 (0.012) | 0.258 (0.012) | 0.037 (0.013)
  Week 16 | 0.235 (0.012) | 0.242 (0.012) | 0.026 (0.013)
  Week 24 | 0.222 (0.012) | 0.245 (0.012) | 0.024 (0.013)
  Week 32 | 0.198 (0.013) | 0.241 (0.013) | 0.018 (0.013)
  Week 40 | 0.197 (0.012) | 0.206 (0.012) | -0.000 (0.012)
  Week 48 | 0.181 (0.013) | 0.210 (0.013) | -0.002 (0.013)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry, centre and baseline value; Mean Difference (Final Values) = 0.183, Standard Error of Mean 0.018 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry, centre and baseline value; Mean Difference (Final Values) = 0.212, Standard Error of Mean 0.018 — Tiotropium Respimat 10mcg - Placebo

50. Secondary Outcome: Change From Baseline in FVC AUC0-3 After 2, 8, 16, 24, 32, 40 and 48 Weeks
Description: FVC AUC0-3 represents the Area under Curve over the time interval from 0 to 3 hours after 2, 8, 16, 24, 32, 40 and 48 weeks. The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: as for outcome 1
Population: Full Analysis Set - Clinic Spirometry (FAS-PFT)
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 324 | 324 | 307
Litres
  Week 2 | 0.513 (0.024) | 0.522 (0.024) | 0.140 (0.025)
  Week 8 | 0.463 (0.026) | 0.521 (0.026) | 0.117 (0.027)
  Week 16 | 0.466 (0.026) | 0.488 (0.026) | 0.108 (0.027)
  Week 24 | 0.468 (0.027) | 0.498 (0.027) | 0.092 (0.027)
  Week 32 | 0.438 (0.027) | 0.477 (0.027) | 0.075 (0.028)
  Week 40 | 0.417 (0.027) | 0.406 (0.027) | 0.029 (0.028)
  Week 48 | 0.387 (0.028) | 0.411 (0.028) | 0.018 (0.029)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry, centre and baseline value; Mean Difference (Final Values) = 0.369, Standard Error of Mean 0.040 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry, centre and baseline value; Mean Difference (Final Values) = 0.393, Standard Error of Mean 0.040 — Tiotropium Respimat 10mcg - Placebo

51. Secondary Outcome: Weekly Mean Morning Pre-dose PEFRs
Description: Weekly mean morning pre-dose peak expiratory flow rates (PEFRs). The means are adjusted for centre, smoking status at entry, and baseline value.
Time Frame: Weeks 2, 8, 16, 24, 32, 40, 48
Population: Full Analysis Set - Diary (FAS-DRY)
Measure: Mean (Standard Error); unit: Litres/minute
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 322 | 324 | 308
Litres/minute
  Week 2 | 245.7 (1.6) | 245.4 (1.6) | 226.9 (1.6)
  Week 8 | 252.4 (2.3) | 253.9 (2.3) | 229.4 (2.4)
  Week 16 | 257.5 (2.8) | 258.4 (2.8) | 231.6 (2.9)
  Week 24 | 260.5 (3.2) | 263.8 (3.2) | 230.9 (3.2)
  Week 32 | 261.5 (3.2) | 264.6 (3.2) | 232.6 (3.3)
  Week 40 | 260.7 (3.2) | 264.7 (3.2) | 231.1 (3.3)
  Week 48 | 260.3 (3.4) | 264.1 (3.4) | 232.4 (3.5)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, centre,smoking status at entry and baseline value; Mean Difference (Final Values) = 27.9, Standard Error of Mean 4.9 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, centre,smoking status at entry and baseline value; Mean Difference (Final Values) = 31.7, Standard Error of Mean 4.9 — Tiotropium Respimat 10mcg - Placebo

52. Secondary Outcome: Weekly Mean Morning Evening PEFRs
Description: Weekly mean evening peak expiratory flow rates (PEFRs). The means are adjusted for centre, smoking status at entry, and baseline value.
Time Frame: Weeks 2, 8, 16, 24, 32, 40, 48
Population: Full Analysis Set - Diary (FAS-DRY)
Measure: Mean (Standard Error); unit: Litres/minute
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 319 | 322 | 309
Litres/minute
  Week 2 | 262.7 (1.7) | 265.0 (1.7) | 237.5 (1.7)
  Week 8 | 267.9 (2.5) | 273.5 (2.5) | 240.6 (2.5)
  Week 16 | 272.7 (3.0) | 276.3 (3.0) | 240.8 (3.1)
  Week 24 | 275.5 (3.2) | 280.3 (3.2) | 241.9 (3.3)
  Week 32 | 276.6 (3.3) | 279.7 (3.2) | 241.0 (3.3)
  Week 40 | 274.0 (3.3) | 280.5 (3.2) | 240.5 (3.2)
  Week 48 | 274.0 (3.4) | 281.0 (3.4) | 241.9 (3.5)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, centre,smoking status at entry and baseline value; Mean Difference (Final Values) = 32.0, Standard Error of Mean 4.9 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, centre,smoking status at entry and baseline value; Mean Difference (Final Values) = 39.1, Standard Error of Mean 4.9 — Tiotropium Respimat 10mcg - Placebo

53. Secondary Outcome: Weekly Mean Number of Puffs of Rescue Medication Per Day
Description: Weekly mean number of puffs of rescue medication used per day as required (PRN salbutamol). The means are adjusted for centre, smoking status at entry, and baseline value.
Time Frame: Weeks 2, 8, 16, 24, 32, 40, 48
Population: Full Analysis Set - Diary (FAS-DRY)
Measure: Mean (Standard Error); unit: Puffs
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 321 | 324 | 311
Puffs
  Week 2 | 2.0 (0.1) | 2.0 (0.1) | 2.8 (0.1)
  Week 8 | 2.3 (0.1) | 2.0 (0.1) | 3.0 (0.1)
  Week 16 | 2.5 (0.1) | 2.1 (0.1) | 3.0 (0.1)
  Week 24 | 2.5 (0.1) | 2.3 (0.1) | 3.0 (0.1)
  Week 32 | 2.7 (0.1) | 2.3 (0.1) | 3.1 (0.1)
  Week 40 | 2.7 (0.1) | 2.4 (0.1) | 3.2 (0.1)
  Week 48 | 2.8 (0.1) | 2.5 (0.1) | 3.2 (0.1)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p = 0.0169, ANCOVA; ANCOVA analysis with terms for treatment, centre,smoking status at entry and baseline value; Mean Difference (Final Values) = -0.4, Standard Error of Mean 0.2 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, centre,smoking status at entry and baseline value; Mean Difference (Final Values) = -0.7, Standard Error of Mean 0.2 — Tiotropium Respimat 10mcg - Placebo

54. Secondary Outcome: Mahler TDI Scores
Description: Mahler Transitional Dyspnoea Index (TDI) scores measured as change in functional impairment, change in magnitude of tasks and change in magnitude of efforts over the treatment period. The means are adjusted for centre, smoking status at entry and baseline value.
  Worst score = -3, best score = +3
Time Frame: Week 48
Population: Full Analysis Set - Transitional Dyspnoea Index (FAS-TDI)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 310 | 305 | 279
Points on a scale
  Functional Impairment | 0.630 (0.057) | 0.577 (0.057) | 0.318 (0.060)
  Magnitude of Task | 0.654 (0.057) | 0.621 (0.057) | 0.275 (0.060)
  Magnitude of Effort | 0.604 (0.061) | 0.594 (0.062) | 0.264 (0.065)

55. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Scores
Description: Saint George's Respiratory Questionnaire (SGRQ) Scores impacts, activities and symptoms. Worst score = 100, best score = 0.
  The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: Week 48
Population: Full Analysis Set - Saint George's Respiratory Questionnaire (FAS-QOL)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 310 | 304 | 276
Points on a scale
  Symptoms | 40.680 (1.116) | 42.108 (1.128) | 48.244 (1.185)
  Activities | 58.529 (0.897) | 57.045 (0.906) | 60.921 (0.953)
  Impacts | 28.858 (0.783) | 29.532 (0.791) | 32.239 (0.832)

56. Secondary Outcome: COPD Symptoms Scores
Description: COPD symptoms Scores - wheezing, shortness of breath, coughing and tightness of chest over the treatment period.
  Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: Week 48
Population: Full Analysis Set - COPD symptoms (FAS-SYM)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 325 | 324 | 304
Points on a scale
  Wheezing | 0.66 (0.04) | 0.72 (0.04) | 0.85 (0.04)
  Shortness of Breath | 1.42 (0.04) | 1.41 (0.04) | 1.61 (0.04)
  Coughing | 0.96 (0.04) | 1.05 (0.04) | 1.06 (0.04)
  Tightness of Chest | 0.51 (0.04) | 0.55 (0.04) | 0.64 (0.04)

57. Secondary Outcome: PGE Scores
Description: Physician's Global evaluation (PGE) scores over the treatment period. Scale: 1-2 = Poor, 3-4 = Fair, 5-6 = Good, 7-8 = Excellent The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: Week 48
Population: Full Analysis Set - Physician's Global Evaluation (FAS-PGE)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 324 | 325 | 305
Points on a scale | 4.90 (0.06) | 4.84 (0.06) | 4.44 (0.06)

58. Secondary Outcome: PGR Scores
Description: Patient's Global rating (PGR) scores over the treatment period. Scale: 1=much better to 7=much worse The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: Week 48
Population: Full Analysis Set - Patient's Global Rating (FAS-PGR)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 312 | 307 | 281
Points on a scale | 2.88 (0.08) | 2.94 (0.08) | 3.42 (0.08)

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after last drug administration.
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 63 | 72 | 56
Other Adverse Events (participants affected / at risk) | 177 | 174 | 182
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Acute coronary syndrome (Cardiac disorders) | 0/338 | 1/335 | 0/334
Angina pectoris (Cardiac disorders) | 0/338 | 2/335 | 0/334
Angina unstable (Cardiac disorders) | 1/338 | 3/335 | 0/334
Arrhythmia (Cardiac disorders) | 1/338 | 0/335 | 0/334
Atrial fibrillation (Cardiac disorders) | 3/338 | 0/335 | 0/334
Atrial flutter (Cardiac disorders) | 0/338 | 0/335 | 1/334
Atrioventricular block (Cardiac disorders) | 0/338 | 1/335 | 0/334
Cardiac failure (Cardiac disorders) | 1/338 | 1/335 | 3/334
Cardiac failure congestive (Cardiac disorders) | 1/338 | 1/335 | 0/334
Coronary artery disease (Cardiac disorders) | 1/338 | 0/335 | 0/334
Myocardial infarction (Cardiac disorders) | 1/338 | 1/335 | 2/334
Myocardial ischaemia (Cardiac disorders) | 0/338 | 0/335 | 1/334
Pericardial effusion (Cardiac disorders) | 1/338 | 0/335 | 0/334
Right ventricular failure (Cardiac disorders) | 1/338 | 0/335 | 1/334
Sick sinus syndrome (Cardiac disorders) | 1/338 | 0/335 | 0/334
Silent myocardial infarction (Cardiac disorders) | 0/338 | 0/335 | 1/334
Supraventricular tachycardia (Cardiac disorders) | 0/338 | 0/335 | 1/334
Vertigo (Ear and labyrinth disorders) | 0/338 | 0/335 | 1/334
Abdominal pain (Gastrointestinal disorders) | 3/338 | 0/335 | 0/334
Abdominal pain upper (Gastrointestinal disorders) | 1/338 | 0/335 | 0/334
Constipation (Gastrointestinal disorders) | 0/338 | 1/335 | 0/334
Diverticulum (Gastrointestinal disorders) | 1/338 | 1/335 | 0/334
Duodenitis (Gastrointestinal disorders) | 0/338 | 0/335 | 1/334
Gastric ulcer (Gastrointestinal disorders) | 0/338 | 0/335 | 1/334
Gastritis (Gastrointestinal disorders) | 0/338 | 0/335 | 2/334
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/338 | 1/335 | 0/334
Hernial eventration (Gastrointestinal disorders) | 0/338 | 1/335 | 0/334
Inguinal hernia (Gastrointestinal disorders) | 1/338 | 0/335 | 0/334
Intestinal obstruction (Gastrointestinal disorders) | 0/338 | 1/335 | 0/334
Intestinal perforation (Gastrointestinal disorders) | 1/338 | 0/335 | 0/334
Jejunal ulcer (Gastrointestinal disorders) | 0/338 | 1/335 | 0/334
Nausea (Gastrointestinal disorders) | 2/338 | 0/335 | 0/334
Neurogenic bowel (Gastrointestinal disorders) | 0/338 | 1/335 | 0/334
Oesophageal stenosis (Gastrointestinal disorders) | 1/338 | 0/335 | 0/334
Peritonitis (Gastrointestinal disorders) | 0/338 | 1/335 | 0/334
Umbilical hernia (Gastrointestinal disorders) | 0/338 | 1/335 | 0/334
Vomiting (Gastrointestinal disorders) | 1/338 | 0/335 | 0/334
Chest pain (General disorders) | 4/338 | 0/335 | 0/334
Death (General disorders) | 0/338 | 1/335 | 0/334
Malaise (General disorders) | 0/338 | 0/335 | 1/334
Pyrexia (General disorders) | 0/338 | 0/335 | 1/334
Cholecystitis (Hepatobiliary disorders) | 1/338 | 0/335 | 0/334
Cholecystitis acute (Hepatobiliary disorders) | 2/338 | 1/335 | 0/334
Biliary sepsis (Infections and infestations) | 0/338 | 1/335 | 0/334
Bronchitis acute (Infections and infestations) | 0/338 | 2/335 | 1/334
Bronchopneumonia (Infections and infestations) | 1/338 | 1/335 | 0/334
Gastroenteritis (Infections and infestations) | 1/338 | 0/335 | 1/334
Influenza (Infections and infestations) | 1/338 | 0/335 | 0/334
Lobar pneumonia (Infections and infestations) | 0/338 | 1/335 | 1/334
Lower respiratory tract infection (Infections and infestations) | 1/338 | 1/335 | 0/334
Pneumonia (Infections and infestations) | 6/338 | 4/335 | 3/334
Pneumonia pneumococcal (Infections and infestations) | 0/338 | 1/335 | 0/334
Pyelonephritis acute (Infections and infestations) | 1/338 | 0/335 | 0/334
Rectal abscess (Infections and infestations) | 1/338 | 0/335 | 0/334
Respiratory tract infection (Infections and infestations) | 1/338 | 0/335 | 1/334
Sepsis (Infections and infestations) | 0/338 | 0/335 | 1/334
Sinusitis (Infections and infestations) | 1/338 | 0/335 | 0/334
Tracheobronchitis (Infections and infestations) | 0/338 | 0/335 | 1/334
Urinary tract infection (Infections and infestations) | 0/338 | 0/335 | 1/334
Viral infection (Infections and infestations) | 0/338 | 0/335 | 1/334
Viral upper respiratory tract infection (Infections and infestations) | 0/338 | 0/335 | 1/334
Wound infection (Infections and infestations) | 0/338 | 1/335 | 0/334
Ankle fracture (Injury, poisoning and procedural complications) | 1/338 | 0/335 | 0/334
Clavicle fracture (Injury, poisoning and procedural complications) | 0/338 | 1/335 | 0/334
Concussion (Injury, poisoning and procedural complications) | 1/338 | 0/335 | 0/334
Contusion (Injury, poisoning and procedural complications) | 0/338 | 2/335 | 0/334
Excoriation (Injury, poisoning and procedural complications) | 0/338 | 1/335 | 0/334
Fall (Injury, poisoning and procedural complications) | 1/338 | 1/335 | 0/334
Graft thrombosis (Injury, poisoning and procedural complications) | 0/338 | 1/335 | 0/334
Humerus fracture (Injury, poisoning and procedural complications) | 0/338 | 0/335 | 1/334
Pubic rami fracture (Injury, poisoning and procedural complications) | 0/338 | 1/335 | 0/334
Road traffic accident (Injury, poisoning and procedural complications) | 0/338 | 1/335 | 0/334
Tendon rupture (Injury, poisoning and procedural complications) | 1/338 | 1/335 | 0/334
Upper limb fracture (Injury, poisoning and procedural complications) | 0/338 | 1/335 | 0/334
Heart rate irregular (Investigations) | 1/338 | 0/335 | 0/334
Liver function test abnormal (Investigations) | 0/338 | 1/335 | 0/334
Hyperglycaemia (Metabolism and nutrition disorders) | 0/338 | 0/335 | 1/334
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/338 | 1/335 | 0/334
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0/338 | 0/335 | 1/334
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0/338 | 1/335 | 0/334
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/338 | 1/335 | 0/334
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1/338 | 0/335 | 0/334
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/338 | 0/335 | 0/334
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/338 | 0/335 | 0/334
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/338 | 1/335 | 0/334
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/338 | 2/335 | 2/334
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/338 | 0/335 | 1/334
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/338 | 0/335 | 0/334
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/338 | 0/335 | 1/334
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/338 | 0/335 | 0/334
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/338 | 2/335 | 1/334
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/338 | 1/335 | 0/334
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/338 | 0/335 | 0/334
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/338 | 1/335 | 0/334
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/338 | 0/335 | 1/334
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/338 | 1/335 | 0/334
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/338 | 1/335 | 0/334
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/338 | 0/335 | 0/334
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/338 | 1/335 | 1/334
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/338 | 1/335 | 0/334
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/338 | 0/335 | 0/334
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/338 | 1/335 | 0/334
Amnesia (Nervous system disorders) | 1/338 | 0/335 | 0/334
Cerebrovascular accident (Nervous system disorders) | 0/338 | 1/335 | 0/334
Ischaemic cerebral infarction (Nervous system disorders) | 0/338 | 1/335 | 0/334
Ischaemic stroke (Nervous system disorders) | 0/338 | 0/335 | 1/334
Loss of consciousness (Nervous system disorders) | 1/338 | 0/335 | 0/334
Paraplegia (Nervous system disorders) | 0/338 | 1/335 | 0/334
Sciatica (Nervous system disorders) | 1/338 | 0/335 | 0/334
Temporal lobe epilepsy (Nervous system disorders) | 1/338 | 0/335 | 0/334
Transient ischaemic attack (Nervous system disorders) | 0/338 | 1/335 | 0/334
Alcoholism (Psychiatric disorders) | 2/338 | 0/335 | 0/334
Completed suicide (Psychiatric disorders) | 1/338 | 0/335 | 0/334
Depression (Psychiatric disorders) | 1/338 | 0/335 | 0/334
Drug dependence (Psychiatric disorders) | 1/338 | 0/335 | 0/334
Tension (Psychiatric disorders) | 1/338 | 0/335 | 0/334
Azotaemia (Renal and urinary disorders) | 0/338 | 1/335 | 0/334
Calculus ureteric (Renal and urinary disorders) | 0/338 | 1/335 | 0/334
Calculus urinary (Renal and urinary disorders) | 0/338 | 0/335 | 1/334
Dysuria (Renal and urinary disorders) | 1/338 | 0/335 | 0/334
Nephropathy toxic (Renal and urinary disorders) | 0/338 | 0/335 | 1/334
Neurogenic bladder (Renal and urinary disorders) | 0/338 | 1/335 | 0/334
Renal failure (Renal and urinary disorders) | 0/338 | 0/335 | 1/334
Renal failure acute (Renal and urinary disorders) | 1/338 | 0/335 | 0/334
Urethral meatus stenosis (Renal and urinary disorders) | 0/338 | 0/335 | 1/334
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/338 | 0/335 | 1/334
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0/338 | 0/335 | 1/334
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 19/338 | 29/335 | 20/334
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/338 | 0/335 | 0/334
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/338 | 0/335 | 0/334
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0/338 | 0/335 | 1/334
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0/338 | 0/335 | 2/334
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0/338 | 0/335 | 1/334
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0/338 | 0/335 | 2/334
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3/338 | 0/335 | 1/334
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2/338 | 1/335 | 2/334
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1/338 | 0/335 | 0/334
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0/338 | 0/335 | 1/334
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0/338 | 0/335 | 1/334
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1/338 | 0/335 | 0/334
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0/338 | 0/335 | 1/334
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/338 | 0/335 | 1/334
Snoring (Respiratory, thoracic and mediastinal disorders) | 0/338 | 0/335 | 1/334
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1/338 | 0/335 | 0/334
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0/338 | 1/335 | 0/334
Postoperative care (Surgical and medical procedures) | 0/338 | 0/335 | 1/334
Transurethral prostatectomy (Surgical and medical procedures) | 0/338 | 0/335 | 1/334
Aortic aneurysm (Vascular disorders) | 0/338 | 1/335 | 1/334
Aortic aneurysm rupture (Vascular disorders) | 0/338 | 1/335 | 0/334
Aortic rupture (Vascular disorders) | 0/338 | 1/335 | 0/334
Deep vein thrombosis (Vascular disorders) | 0/338 | 0/335 | 1/334
Femoral arterial stenosis (Vascular disorders) | 0/338 | 1/335 | 0/334
Hypotension (Vascular disorders) | 0/338 | 1/335 | 0/334
Iliac artery stenosis (Vascular disorders) | 1/338 | 0/335 | 0/334
Peripheral ischaemia (Vascular disorders) | 0/338 | 1/335 | 0/334
Peripheral vascular disorder (Vascular disorders) | 1/338 | 0/335 | 0/334
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Dry mouth (Gastrointestinal disorders) | 25/338 | 44/335 | 7/334
Influenza (Infections and infestations) | 13/338 | 15/335 | 17/334
Nasopharyngitis (Infections and infestations) | 53/338 | 33/335 | 24/334
Upper respiratory tract infection (Infections and infestations) | 17/338 | 17/335 | 19/334
Headache (Nervous system disorders) | 19/338 | 16/335 | 15/334
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 103/338 | 96/335 | 141/334
Cough (Respiratory, thoracic and mediastinal disorders) | 19/338 | 25/335 | 11/334
Pharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19/338 | 17/335 | 9/334

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.